CLINICAL TRIAL: NCT00230919
Title: Weight Loss and Changes in Cardiovascular Risk Markers With a Low Glycemic Load Diet Compared With a Standard National Nutrition Council-recommended Diet: a Randomized Trial
Brief Title: Weight Loss and Changes in Cardiovascular Risk Markers With a Low Glycemic Diet Compared With a Standard Diet
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ullevaal University Hospital (Other)
Collaborators: Norges Forskningsråd, Stenberggata 26, pb. 2700, N-0131 Oslo, Norway (Unknown)
Responsible Party: Department of preventive Cardiology, Ullevaal University Hospital
Organization: Oslo University Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 161327/V50
Record Dates: First submitted 2005-09-30; First posted 2005-10-03 (Estimated); Last update posted 2011-07-01 (Estimated); Status verified 2004-02

CONDITIONS: Obesity; Metabolic Syndrome
Keywords: Obesity,; weight loss,; diet counseling; low-glycemic load
MeSH Terms: conditions — Obesity; Metabolic Syndrome; Weight Loss

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Behavioral: Diet counseling

SUMMARY:
Overweight and obesity is increasing in most countries, including Norway, and the optimal diet for reducing weight is under discussion. The present study in overweight and moderate obese individuals compares a low glycemic load diet with a standard low-fat diet (as recommended from the National Nutrition Council) in an open, randomized trial over 12 months, with changes in weight loss and changes in cardiovascular risk markers as endpoints.

DETAILED DESCRIPTION:
Overweight and obesity is rapidly increasing in most countries, including Norway, and at present there is controversy regarding what diet should be recommended for reducing weight and the complications of obesity.

The present study is performed in in 200 overweight and moderate obese individuals, that is in men with body mass index (BMI) from 28 to 40, and women with BMI 28-35. To be included, the participants should also have at least one component of the metabolic syndrome.

After a medical examination and check for inclusion and exclusion criteria, the participants are randomized to one the two following diets: 1) A low-glycemic load diet aiming at a macronutrient composition with 25-30% of energy from protein, 35-40% from fat and 30-35% from carbohydrate or 2) A low-fat diet aiming at a macronutrient composition with 15% of energy from protein, 25-30% from fat and 55-60% from carbohydrate.

Each group will have 9 dietary counselling sessions in the course of the study; baseline, week 2, month 1,3,4,5,6 and 9. Recommended total energy intake will be individualized based on the metabolic rate at rest for each subject, and using a physical activity level of 1,4. A 500 kcal/day deficit relative to the daily energy requirements will be recommended.

The primary objective will be to compare the effects of the two different diet recommendations with respect to the one-year change in body weight.

As secondary objectives the study will compare the consequences of the two strategies with respect to 3, 6, and 12 months development of the variables glucose/insulin, insulin sensitivity index, number of metabolic syndrome factors, high sensitive C-reactive protein, lipids, lipoprotein B and anthropometric indices (waist /hip ratio). Serum will be frozen for additional parameters as leptin, adiponectin, ghrelin and ICAM. Also to be studied is an additional weight at 18 months follow-up, when no more advice is given past the 9-month visit.

ELIGIBILITY:
Inclusion Criteria:

* Men or women age 30-65,
* BMI in the range 28-35 kg/m2 for women and 28-40kg/m2 for men.
* At least one of the following components of the metabolic syndrome; fasting triglycerides > 1,7, fasting glucose 6,0-6,9, HDL-cholesterol <1,03 (males) or <1,29 (females), Blood pressure >130/85 (with or without treatment), diet-treated diabetes mellitus or drug treated hypertension.
* Stable weight range of 4 kg or less the last 12 weeks,
* No major change in physical activity the last 12 weeks

Exclusion Criteria:

* Any symptomatic cardiovascular disease
* Diabetes requiring drug treatment
* Currently on special diet
* Hepatic/renal dysfunction
* Hypothyroidism (unstable)
* GI disorder impairing compliance with diet recommendation,
* History of unstable psychiatric or medical disorder,
* Need of lipid lowering drug,
* Alcohol or drug abuse,
* Participation in drug trial the last 30 days,
* Use of drugs for weight reduction last 12 weeks, pregnancy or planned pregnancy,
* Obesity of known endocrine origin, history of obesity surgery,
* Uncontrolled hypertension (>160/100),
* Previous participation in >3 weight reduction programs, or within last 12 months,
* Not willing to be randomized,
* Individual judged to be unable to follow instructions and procedures of the study

Ages: 30 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200
Dates: Start 2004-04; Primary Completion 2006-06 (Actual); Study Completion 2006-11 (Actual)

PRIMARY OUTCOMES:
The primary objective will be to compare the effects of the two different diet recommendations with respect to the one-year change in body weight.

SECONDARY OUTCOMES:
Compare the consequences of the two strategies with respect to 3, 6, and 12 months development of the variables; glucose/insulin,
insulin sensitivity index,
number of metabolic syndrome factors,
high sensitive C-reactive protein,
lipids and lipoprotein B and
anthropometric indices (waist /hip ratio)
Fat cell hormones (leptin, adiponectin, ghrelin)
Inflammation markers (ICAM).
Weight at 18 months follow-up.

CONTACTS AND LOCATIONS:
Overall Officials: Tor Ole Klemsdal, MD, Ph.D, Principal Investigator — Ullevaal University Hospital, preventive medicine clinic; Serena Tonstad, MD, Ph.D, Study Chair — Ullevaal University Hospital, preventive medicine clinic
Locations (1):
- Ulleval University Hospital, dep. of preventive cardiology, Oslo, Oslo County, Norway

REFERENCES:
- [Result] Klemsdal TO, Holme I, Nerland H, Pedersen TR, Tonstad S. Effects of a low glycemic load diet versus a low-fat diet in subjects with and without the metabolic syndrome. Nutr Metab Cardiovasc Dis. 2010 Mar;20(3):195-201. doi: 10.1016/j.numecd.2009.03.010. Epub 2009 Jun 6. PMID 19502017
- [Derived] Heggen E, Klemsdal TO, Haugen F, Holme I, Tonstad S. Effect of a low-fat versus a low-gycemic-load diet on inflammatory biomarker and adipokine concentrations. Metab Syndr Relat Disord. 2012 Dec;10(6):437-42. doi: 10.1089/met.2012.0012. Epub 2012 Aug 13. PMID 22889406